CLINICAL TRIAL: NCT01212835
Title: The Use of a Silastic Ring in Open Gastric Bypass for Morbid Obesity and Its Association With Gastroesophageal Reflux Disease
Brief Title: Effect of RING on Gastroesophageal Reflux (GERD) After RYGBP
Acronym: RING
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of follow up
Sponsor: Clinica Gastrobese (Other)
Responsible Party: Principal Investigator, Carlos AS Madalosso, Carlos AS Madalosso, Clinica Gastrobese
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GASTROBESE 005
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Morbid Obesity; Gastroesophageal Reflux Disease; Vomiting
Keywords: Obesity; gastroesophageal reflux disease; Morbid obesity; esophagitis; GERD; silastic ring; Gastric bypass
MeSH Terms: conditions — Obesity, Morbid; Gastroesophageal Reflux; Vomiting; Obesity; Esophagitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- no ring (Sham Comparator): Patients at this group will have RING REMOVED AT THE END OF SURGERY.
  Interventions: Procedure: Sham Comparator: no ring
- RYGBP-Ring (Active Comparator): Open Roux-en-Y gastric bypass with a silastic ring which is performed with linear cut stapler 100 mm and a biliopancreatic limb of 60 cm long and a alimentary limb of 100 cm long. All patients will have a 6.5 cm silastic ring located at the middle of the pouch above of the gastroenteroanastomosis.
  Interventions: Procedure: RYGBP-RING

INTERVENTIONS:
Procedure: Sham Comparator: no ring — Open roux-en-Y gastric bypass not banded
  Arms: no ring
Procedure: RYGBP-RING — Vertical Roux-en-Y banded gastric bypass
  Arms: RYGBP-Ring

SUMMARY:
Silastic rings have been used around the gastric pouch in order to promote better weight loss after Roux-and-Y gastric bypass surgery ( RYGBP). However the investigators have shown that some patients developed gastroesophageal reflux disease after RYGBP in a previous study. The investigators hypothesized that the use of a silastic ring may play a role in promoting GERD after this operation.

DETAILED DESCRIPTION:
This is a randomized controlled double blind trial designed to identify if the use of the ring induces food intolerance and vomiting which may lead a esophageal mucosal erosions and/or GERD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Indications for bariatric surgery (BMI over 40Kg/m2 or over 35Kg/m2 associated to a life-treating morbid conditions.
* Acceptance to be submitted to a 24h pH-monitoring and esophageal manometry
* No contra-indication for gastric bypass
* Absence of previous gastric surgery
* Option for open gastric bypass

Exclusion Criteria:

* Inferior and superior total teeth prosthesis
* Poor surgical conditions

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Occurence of gastroesophageal reflux disease | march 2010 to march 2014
  Patients are intra-operatively selected to receive or not a silastic ring following a open gastric bypass. These patients will be evaluated for GERD with upper endoscopy, 24h ph-monitoring, validated questionnaires which will be performed at 6 month, 1 and 2 years.

SECONDARY OUTCOMES:
The role of the ring in open GBP in terms of weight loss | march 2010 to march 2014
  It will be possible to evaluate the weight loss among the groups: 1) with ring and, 2) without a ring
The impact of the ring on food tolerance | March 2010 to March 2014
  To identify food intolerance among the groups: 1) with the ring, and 2) without the ring.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Navarini, M.D., Study Chair — Clinica Gastrobese; Carlos AS Madalosso, M.D., Principal Investigator — Clinica Gastrobese; Iran Moraes Jr, M.D., Study Chair — Clinica Gastrobese; Fabio R Barao, Admn, Study Director — Protocol control
Locations (3):
- Brazil (3):
  - Clínica Gastrobese, Passo Fundo, Rio Grande do Sul
  - Gastrobese Clinic, Passo Fundo, Rio Grande do Sul
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul

REFERENCES:
- [Result] Madalosso CA, Gurski RR, Callegari-Jacques SM, Navarini D, Thiesen V, Fornari F. The impact of gastric bypass on gastroesophageal reflux disease in patients with morbid obesity: a prospective study based on the Montreal Consensus. Ann Surg. 2010 Feb;251(2):244-8. doi: 10.1097/SLA.0b013e3181bdff20. PMID 20010088